CLINICAL TRIAL: NCT03546621
Title: A Multicenter, Open-label, Randomized Clinical Study to Assess Efficacy and Safety of 3 Doses of Myrcludex B for 24 Weeks in Combination With Tenofovir Compared to Tenofovir Alone to Suppress HBV Replication in Patients With Chronic Hepatitis D
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hepatera Ltd. (Industry)
Collaborators: Data Matrix Solutions (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MYR 202
Record Dates: First submitted 2018-05-23; First posted 2018-06-06 (Actual); Results first posted 2019-12-30 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-04

CONDITIONS: Chronic Hepatitis D Infection With Hepatitis B
Keywords: Hepatitis D
MeSH Terms: conditions — Hepatitis D | interventions — myrcludex-B; Tenofovir

STUDY DESIGN:
Intervention Model Description: Multicenter, Open-label, Randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm A (Experimental): Myrcludex B, 2 mg/day subcutaneously (s.c.) for 24 weeks + tenofovir with a further follow-up period of 24 weeks of continued tenofovir therapy.
  Interventions: Drug: Myrcludex B; Drug: Tenofovir
- Arm B (Experimental): Myrcludex B, 5 mg/day subcutaneously (s.c.) for 24 weeks + tenofovir with a further follow-up period of 24 weeks of continued tenofovir therapy.
  Interventions: Drug: Myrcludex-B; Drug: Tenofovir
- Arm C (Experimental): Myrcludex B, 10 mg/day subcutaneously (s.c.) for 24 weeks + tenofovir with a further follow-up period of 24 weeks of continued tenofovir therapy.
  Interventions: Drug: Myrcludex-B; Drug: Tenofovir
- Arm D (Active Comparator): tenofovir treatment for 48 weeks
  Interventions: Drug: Tenofovir

INTERVENTIONS:
Drug: Myrcludex B — 2 mg, once daily, subcutaneously
  Arms: Arm A
Drug: Myrcludex-B — 5 mg, once daily, subcutaneously
  Arms: Arm B
Drug: Myrcludex-B — 10 mg, once daily, subcutaneously
  Arms: Arm C
Drug: Tenofovir — tenofovir disoproxil 245 mg, equivalent to tenofovir disoproxil fumarate 300 mg
  Other Names: Viread

SUMMARY:
This is a multicenter, open-label, randomized clinical trial to Assess Efficacy and Safety of 3 Doses of Myrcludex B for 24 Weeks in Combination with Tenofovir Compared to Tenofovir Alone to Suppress HBV Replication in Patients with Chronic Hepatitis D

DETAILED DESCRIPTION:
This is a multicenter, open-label, randomised, phase II study.

The study will be conducted in Russia and Germany. The study is designed to evaluate the benefit of 3 MXB doses versus observation in patients on background therapy with tenofovir, suffering from hepatitis delta with very limited therapeutic options; the patients will be randomized 1:1:1:1 into 3 treatment arms and an observation arm. Patients with compensated cirrhosis at screening will be stratified to allow similar distribution into each treatment arm. If patients were not receiving treatment with nucleoside/nucelotide analogue, the comparator/background drug will be initiated after the eligibility confirmation, for 12 weeks prior to randomization visit; patients who previously received tenofovir will continue the dosing; patients on different nucleoside/nucleotide analogue will be switched to tenofovir. Observation is considered an adequate control group, as daily placebo injections for 24 weeks are regarded not feasible and ethically questionable.

It is planned to screen 200 patients, and 120 patients will be randomised into four treatment arms in the 1:1:1:1 ratio.

* Arm A (30 patients): Myrcludex B, 2 mg/day subcutaneously (s.c.) for 24 weeks + tenofovir with a further follow-up period of 24 weeks of continued tenofovir therapy.
* Arm B (30 patients): Myrcludex B, 5 mg/day subcutaneously (s.c.) for 24 weeks + tenofovir with a further follow-up period of 24 weeks of continued tenofovir therapy.
* Arm C (30 patients): Myrcludex B, 10 mg/day subcutaneously (s.c.) for 24 weeks + tenofovir with a further follow-up period of 24 weeks of continued tenofovir therapy.
* Arm D (30 patients): tenofovir treatment for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 65 years inclusively at the time of signing Informed Consent Form.
2. Positive serum HBsAg for at least 6 months before Screening.
3. Positive serum anti-HDV antibody for at least 6 months before screening.
4. Positive PCR results for serum HDV RNA at Screening.
5. Patients with liver cirrhosis, irrespective of previous interferon treatment .
6. Patients without liver cirrhosis, who failed prior interferon treatment or for whom, in the opinion of the Investigator, such treatment is currently contraindicated (including history of interferon intolerance) .
7. Alanine aminotransferase level >1 x ULN, but less than 10 x ULN.
8. Previous nucleotide/nucleoside analogue treatment within at least 12 weeks prior to the planned start of study treatment or subject's willingness to take tenofovir for at least 12 weeks prior to the planned start of study treatment.
9. Negative urine pregnancy test for females of childbearing potential.
10. Inclusion criteria for female subjects:

    * Postmenopausal for at least 2 years, or
    * Surgically sterile (total hysterectomy or bilateral oophorectomy, bilateral tubal ligation, staples, or another type of sterilization), or
    * Abstinence from heterosexual intercourse throughout the study, or
    * Willingness to use highly effective contraception throughout the study and for 3 months after the last dose of the study medication.
11. Male and female subjects must agree to use a highly effective contraception throughout the study and for 3 months after the last dose of the study medication.
12. Male subjects must agree not to donate sperm throughout the study and for 3 months after the last dose of the study medication.

Exclusion Criteria:

1. Child-Pugh score of B-C or over 6 points.
2. HCV or HIV coinfection. Subjects with anti-HCV antibodies can be enrolled, if screening HCV RNA test is negative.
3. Creatinine clearance <60 mL/min.
4. Total bilirubin ≥ 2mg/dL. Patients with higher total bilirubin values may be included after the consultation with the Study's Medical Monitor, if such elevation can be clearly attributed to Gilbert's syndrome associated with low-grade hyperbilirubinemia.
5. Any previous or current malignant neoplasms, including hepatic carcinoma.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-02-16 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heiner Wedemeyer, MD,PhD, Principal Investigator — Dept. of Gastroenterology, Hepatology and Endocrinology Medizinische Hochschule Hannover
Locations (15):
- Germany (4):
  - Ifi-Institut für interdisziplinäre Medizin an der Asklepios Klinik St. Georg, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf Medizinische Klinik Studienambulanz Hepatologie, Hamburg
  - Klinik für Gastroenterologie, Hepatologie und Endokrinologie, Medizinische Hochschule Hannover, Hanover
  - UniversitätsKlinikum Heidelberg - Medizinische Klinik, Abteilung Klinische Pharmakologie & Pharmakoepidemiologie, Heidelberg
- Russia (11):
  - State Budgetary educational institution of higher professional education "South Ural State Medical University" Ministry of healthcare, Chelyabinsk
  - State Autonomous Healthcare Institution "Republican Clinical Infectious Diseases Hospital named after Prof. A.F. Agafonov "(SAHI RCID), Kazan'
  - Federal Budget Institution of Science "Central Research Institute of Epidemiology" of The Federal Service on Customers' Rights Protection and Human Well-being Surveillance, Moscow
  - LLC "Clinic of Modern Medicine", Moscow
  - Moscow Regional Research Clinical Institute n.a. M.F. Vladimirskiy, Moscow
  - State Budget Health Institution of Moscow "Infectious Clinical Hospital No. 1 of the Moscow Healthcare Department", Moscow
  - State Budgetary Healthcare Institution "Moscow Clinical Scientific and Practical Center of the Department of Public Health of Moscow", Moscow
  - State Budgetary Educational Institution of Higher Professional Education "Novosibirsk State Medical University" of the Ministry of Health of the Russian Federation, Novosibirsk
  - Medical Company "Hepatolog", Samara
  - Stavropol Regional Clinical Hospital, Stavropol
  - State Budgetary institution of the Republic of Sakha (Yakutia) "Yakutsk Clinical Hospital", Yakutsk

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Allweiss L, Volmari A, Suri V, Wallin JJ, Flaherty JF, Manuilov D, Downie B, Lutgehetmann M, Bockmann JH, Urban S, Wedemeyer H, Dandri M. Blocking viral entry with bulevirtide reduces the number of HDV-infected hepatocytes in human liver biopsies. J Hepatol. 2024 Jun;80(6):882-891. doi: 10.1016/j.jhep.2024.01.035. Epub 2024 Feb 8. PMID 38340811
- [Derived] Hollnberger J, Liu Y, Xu S, Chang S, Martin R, Manhas S, Aeschbacher T, Han B, Yazdi T, May L, Han D, Shornikov A, Flaherty J, Manuilov D, Suri V, Asselah T, Lampertico P, Wedemeyer H, Aleman S, Richards C, Mateo R, Maiorova E, Cihlar T, Mo H, Urban S. No virologic resistance to bulevirtide monotherapy detected in patients through 24 weeks treatment in phase II and III clinical trials for chronic hepatitis delta. J Hepatol. 2023 Sep;79(3):657-665. doi: 10.1016/j.jhep.2023.04.027. Epub 2023 Apr 27. PMID 37120031
- [Derived] Wedemeyer H, Schoneweis K, Bogomolov P, Blank A, Voronkova N, Stepanova T, Sagalova O, Chulanov V, Osipenko M, Morozov V, Geyvandova N, Sleptsova S, Bakulin IG, Khaertynova I, Rusanova M, Pathil A, Merle U, Bremer B, Allweiss L, Lempp FA, Port K, Haag M, Schwab M, Zur Wiesch JS, Cornberg M, Haefeli WE, Dandri M, Alexandrov A, Urban S. Safety and efficacy of bulevirtide in combination with tenofovir disoproxil fumarate in patients with hepatitis B virus and hepatitis D virus coinfection (MYR202): a multicentre, randomised, parallel-group, open-label, phase 2 trial. Lancet Infect Dis. 2023 Jan;23(1):117-129. doi: 10.1016/S1473-3099(22)00318-8. Epub 2022 Sep 13. PMID 36113537

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 120 randomized patients 118 started treatment with study medication (2 patients from Tenofovir only group withdrew before treatment)
Period: Overall Study
Arm/Group | Arm A | Arm B | Arm C | Arm D
Started | 28 | 32 | 30 | 28 (2 patients from Tenofovir only group withdrew from the study before treatment.)
Completed | 28 | 29 | 28 | 25
Not Completed | 0 | 3 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 1
Not completed — Progressive disease | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Arm C | Arm D | Total
Number analyzed (Participants) | 28 | 32 | 30 | 28 | 118
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 28 | 32 | 30 | 28 | 118
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.4 (8.3) | 40.9 (9.5) | 41.8 (11.3) | 38.5 (8.7) | 40.2 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 7 | 8 | 39
  Male | 15 | 21 | 23 | 20 | 79
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 7 | 1 | 3 | 5 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 21 | 30 | 27 | 23 | 101
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Height (cm) [Mean (Standard Deviation); unit: cm.] | 168.5 (8.3) | 172.9 (7.4) | 173.8 (9.8) | 172.8 (9.4) | 172.0 (8.9)
Body Weight (kg) [Mean (Standard Deviation); unit: kg.] | 70.19 (13.54) | 75.09 (12.54) | 77.59 (13.72) | 79.15 (17.21) | 75.53 (14.49)
Body Mass Index (kg/m²) [Number; unit: participants]
  <30 kg/m² | 27 | 31 | 28 | 22 | 108
  ≥30 kg/m² | 1 | 1 | 2 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: HDV RNA Response at Week 24
Description: HDV RNA negativation or decrease by ≥2 log10 from baseline to Week 24
Time Frame: 24 weeks
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm D
Number analyzed (Participants) | 28 | 32 | 30 | 28
Participants
  Responder | 15 | 16 | 23 | 1
  Non-Responder | 13 | 16 | 7 | 27
Statistical Analysis 1: Comparison: Arm A vs Arm B vs Arm C; For each of the three Myrcludex B treatment groups, a null hypothesis of no clinically significant difference in proportion of responders compared to the control group (Tenofovir only), at week 24, were tested using the one-sided Wald test for superiority, at a one-sided overall significance level of 0.05 adjusted for multiple testing according to Bonferroni-Holm, with the superiority limit (test margin) set to 5%; Test type: Superiority; p < .0001, Bonferroni-Holm

2. Secondary Outcome: Durability of HDV RNA Response
Description: Durability of HDV RNA response to 24 weeks post treatment
Time Frame: 48 weeks
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm D
Number analyzed (Participants) | 28 | 32 | 30 | 28
Participants
  Response at Week 24 only | 15 | 16 | 23 | 1
  Response at Week 24 and 48 | 2 | 1 | 3 | 0
Statistical Analysis 1: Comparison: Arm A vs Arm D; Week 48. Two-sided Fisher's exact tests were used to test null hypothesis of no difference in the proportion of responders compared to the Tenofovir only group. Separate comparisons were made for each of the three Myrcludex B groups versus the control group, and the adjusted p-values were computed using the Bonferroni-Holm method; Test type: Superiority; p = 0.9818, Bonferroni-Holm — A test is considered as statistically significant if the adjusted p-value is smaller than 0.05
Statistical Analysis 2: Comparison: Arm B vs Arm D; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 1.0000, Bonferroni-Holm — A test is considered as statistically significant if the adjusted p-value as smaller than 0.05
Statistical Analysis 3: Comparison: Arm C vs Arm D; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.7132, Bonferroni-Holm — The threshold for statistical significance was p=0.05

3. Secondary Outcome: Combined Response: HDV RNA Response and Normal ALT at Treatment Week 24
Description: Combined response: HDV RNA negativation or ≥2 log decline and normal ALT at treatment week 24
Time Frame: 24 weeks
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm D
Number analyzed (Participants) | 28 | 32 | 30 | 28
Participants
  Week 24: Responder | 6 | 9 | 11 | 0
  Week 24: Non-Responder | 22 | 23 | 19 | 28
  Week 48: Responder | 2 | 1 | 1 | 0
  Week 48: Non-Responder | 26 | 31 | 29 | 28
Statistical Analysis 1: Comparison: Arm A vs Arm D; Fisher's exact test was used to test a null hypothesis of no difference in proportions against a two-sided alternative hypothesis. Separate tests were performed for each of the three Myrcludex B treatment groups against the control group, at week 24 and week 48, and adjusted p-values were computered using the Bonferroni-Holm method. This analysis, and presentation of descriptive statistics, was repeated for the subgroups of patients with normal/abnormal baseline ALT values; Test type: Superiority; p = 0.0232, Bonferroni-Holm — A test is considered as statistically significant if the adjusted p-value is smaller than 0.05
Statistical Analysis 2: Comparison: Arm B vs Arm D; Fisher's exact test was used to test a null hypothesis of no difference in proportions against a two-sided alternative hypothesis. Separate tests were performed for each of the three Myrcludex B treatment groups against the control group, at week 24 and week 48, and adjusted p-values were computered using the Bonferroni-Holm method; Test type: Superiority; p = 0.0047, Bonferroni-Holm — The threshold for statistical significance was p=0.05
Statistical Analysis 3: Comparison: Arm C vs Arm D; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.0010, Bonferroni-Holm — The threshold for statistical significance was p=0.05

4. Secondary Outcome: Changes in ALT Values
Description: Changes in ALT values at Week 24 and Week 48 compared to baseline.
Time Frame: 24 and 48 weeks
Population: mITT
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Arm A | Arm B | Arm C | Arm D
Number analyzed (Participants) | 28 | 32 | 30 | 28
U/L
  Change from Baseline to Week 24: number analyzed (Participants) | 28 | 30 | 29 | 25
  Change from Baseline to Week 24 | -49.6 (58.7) | -79.4 (84.2) | -78.9 (81.1) | -29.2 (61.4)
  Change from Baseline to Week 48: number analyzed (Participants) | 28 | 29 | 29 | 25
  Change from Baseline to Week 48 | -1.6 (72.8) | -18.2 (94.4) | 1.4 (76.0) | -26.3 (39.0)
Statistical Analysis 1: Comparison: Arm A vs Arm D; Week 24. The change from baseline to week 24 and week 48 in ALT levels was performed using van Elteren tests. Fisher's exact test was used to test a null hypothesis of no difference in proportions (of patients with normal ALT values) against a two-sided alternative hypothesis. Separate tests were performed for each of the three Myrcludex B treatment groups against the control group, at week 24 and week 48, and adjusted p-values were computed using the Bonferroni-Holm method; Test type: Superiority; p = 0.1642, Bonferroni-Holm — A test is considered as statistically significant if the adjusted p-value is smaller than 0.05
Statistical Analysis 2: Comparison: Arm B vs Arm D; Week 24; Test type: Superiority; p = 0.0428, Bonferroni-Holm — A test is considered statistically significant if the adjusted p-value is smaller than 0.05
Statistical Analysis 3: Comparison: Arm C vs Arm D; Week 24; Test type: Superiority; p = 0.0428, Bonferroni-Holm — A test is considered statistically significant if the adjusted p-value is smaller than 0.05
Statistical Analysis 4: Comparison: Arm A vs Arm D; Week 48; Test type: Superiority; p = 0.2388, Boferroni-Holm — A test is considered as statistically significant if the adjusted p-value is smaller than 0.05
Statistical Analysis 5: Comparison: Arm B vs Arm D; Week 48; Test type: Superiority; p = 0.7157, Bonferroni-Holm — A test is considered as statistically significant if the adjusted p-value is smaller than 0.05
Statistical Analysis 6: Comparison: Arm C vs Arm D; Week 48; Test type: Superiority; p = 0.2388, Bonferroni-Holm — A test is considered as statistically significant if the adjusted p-value is smaller than 0.05

5. Secondary Outcome: Change (Absence of Increase) in Fibrosis Marker
Description: Change (absence of increase) in fibrosis marker: serum alpha-2-macroglobulin at Week 24 and Week 48 compared to baseline
Time Frame: 24 and 48 weeks
Population: mITT
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Arm A | Arm B | Arm C | Arm D
Number analyzed (Participants) | 28 | 32 | 30 | 28
g/L
  Change from Baseline to Week 24: number analyzed (Participants) | 23 | 23 | 23 | 23
  Change from Baseline to Week 24 | -0.076 (0.320) | 0.020 (0.280) | 0.024 (0.257) | -0.141 (0.607)
  Change from Baseline to Week 48: number analyzed (Participants) | 23 | 22 | 21 | 23
  Change from Baseline to Week 48 | -0.056 (0.416) | 0.075 (0.360) | -0.008 (0.265) | -0.031 (0.485)
Statistical Analysis 1: Comparison: Arm A vs Arm D; Week 24. Two-sided van Elteren tests, stratified by presence of cirrhosis, were used to test for differences compared to the control group. Separate comparisons were made for each of the three MXB groups versus the control group, and adjusted p-values were computed using the Bonferroni-Holm method; Test type: Superiority; p = 0.7416, Bonferroni-Holm — A test is considered as statistically significant if the adjusted p-value is smaller than 0.05
Statistical Analysis 2: Comparison: Arm B vs Arm D; Week 24; Test type: Superiority; p = 0.4434, Bonferroni-Holm — A test is considered as statistically significant if the adjusted p-value is smaller than 0.05
Statistical Analysis 3: Comparison: Arm C vs Arm D; Week 24; Test type: Superiority; p = 0.7371, Bonferroni-Holm — A test is considered as statistically significant if the adjusted p-value is smaller than 0.05
Statistical Analysis 4: Comparison: Arm A vs Arm D; Week 48; Test type: Superiority; p = 1.0000, Bonferroni-Holm — A test is considered as statistically significant if the adjusted p-value is smaller than 0.05
Statistical Analysis 5: Comparison: Arm B vs Arm D; Week 48; Test type: Superiority; p = 0.9441, Bonferroni-Holm — A test is considered as statistically significant if the adjusted p-value is smaller than 0.05
Statistical Analysis 6: Comparison: Arm C vs Arm D; Week 48; Test type: Superiority; p = 1.0000, Bonferroni-Holm — A test is considered as statistically significant if the adjusted p-value is smaller than 0.05

6. Secondary Outcome: Change in Hepatitis B Surface Antigen
Description: Changes in hepatitis B surface antigen (HBsAg) (defined as decline in HBsAg levels, disappearance of HBsAg and HBsAg seroconversion to anti-HBsAg) at week 24 and week 48 compared to baseline
Time Frame: 24 and 48 weeks
Population: mITT
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Arm A | Arm B | Arm C | Arm D
Number analyzed (Participants) | 28 | 32 | 30 | 28
IU/mL
  Change from Baseline to Week 24: number analyzed (Participants) | 27 | 30 | 28 | 25
  Change from Baseline to Week 24 | -0.048 (0.392) | 0.003 (0.175) | 0.034 (0.106) | 0.025 (0.239)
  Change from Baseline to Week 48: number analyzed (Participants) | 27 | 29 | 28 | 24
  Change from Baseline to Week 48 | -0.138 (0.288) | -0.162 (0.412) | -0.134 (0.175) | -0.070 (0.186)
Statistical Analysis 1: Comparison: Arm A vs Arm D; Week 24. The change from baseline to Week 24 in HBsAg was performed using van Elteren tests. Tests were performed on log-10 transformed data. Separare comparisons were made for each of the three Myrcludex B groups versus the control group, and the adjusted values were computed using the Bonferroni-Holm method; Test type: Superiority; p = 0.5984, Bonferroni-Holm — A test is considered as statistically significant if the adjusted p-value is smaller than 0.05; Bonferroni-Holm
Statistical Analysis 2: Comparison: Arm B vs Arm D; Week 24; Test type: Superiority; p = 0.7529, Bonferroni-Holm — A test is considered as statistically significant if the adjusted p-value is smaller than 0.05
Statistical Analysis 3: Comparison: Arm C vs Arm D; Week 24; Test type: Superiority; p = 0.3305, Bonferroni-Holm — A test is considered as statistically significant if the adjusted p-value is smaller than 0.05
Statistical Analysis 4: Comparison: Arm A vs Arm D; Week 48; Test type: Superiority; p = 1.0000, Bonferroni-Holm — A test is considered as statistically significant if the adjusted p-value is smaller than 0.05
Statistical Analysis 5: Comparison: Arm B vs Arm D; Week 48; Test type: Superiority; p = 1.0000, Bonferroni-Holm — A test is considered as statistically significant if the adjusted p-value is smaller than 0.05
Statistical Analysis 6: Comparison: Arm C vs Arm D; Week 48; Test type: Superiority; p = 1.0000, Bonferroni-Holm — A test is considered as statistically significant if the adjusted p-value is smaller than 0.05

7. Secondary Outcome: Change in HBV DNA Levels at Week 24 and Week 48 Compared to Baseline
Description: Change in hepatitis B virus (HBV) DNA levels at Week 24 and Week 48 compared to baseline.
Time Frame: 24 and 48 weeks
Population: mITT
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Arm A | Arm B | Arm C | Arm D
Number analyzed (Participants) | 28 | 32 | 30 | 28
IU/mL
  Change from Baseline to Week 24: number analyzed (Participants) | 27 | 30 | 28 | 25
  Change from Baseline to Week 24 | -0.314 (0.956) | -0.484 (1.106) | -0.173 (1.144) | -0.343 (1.151)
  Change from Baseline to Week 48: number analyzed (Participants) | 27 | 29 | 28 | 24
  Change from Baseline to Week 48 | -0.244 (0.828) | -0.194 (1.416) | -0.267 (1.275) | -0.257 (0.979)
Statistical Analysis 1: Comparison: Arm A vs Arm D; Week 24. Two-sided van Elteren tests, stratified by presence of cirrhosis, were used to test for differences compared to the control group. Tests were performed on log-10 transformed data. Separate comparisons were made for each of the three MXB groups versus the control group, and adjusted p-values were computed using the Bonferroni-Holm method; Test type: Superiority; p = 1.0000, Bonferroni-Holm — A test is considered as statistically significant if the adjusted p-value is smaller than 0.05
Statistical Analysis 2: Comparison: Arm B vs Arm D; Week 24; Test type: Superiority; p = 1.0000, Bonferroni-Holm
Statistical Analysis 3: Comparison: Arm C vs Arm D; Week 24; Test type: Superiority; p = 1.0000, Bonferroni-Holm
Statistical Analysis 4: Comparison: Arm A vs Arm D; Week 48; Test type: Superiority; p = 1.0000, Bonferroni-Holm — A test is considered as statistically significant if the adjusted p-value is smaller than 0.05
Statistical Analysis 5: Comparison: Arm B vs Arm D; Week 48; Test type: Superiority; p = 1.0000, Bonferroni-Holm — A test is considered as statistically significant if the adjusted p-value is smaller than 0.05
Statistical Analysis 6: Comparison: Arm C vs Arm D; Week 48; Test type: Superiority; p = 1.0000, Bonferroni-Holm — A test is considered as statistically significant if the adjusted p-value is smaller than 0.05

8. Secondary Outcome: Absence of a Fibrosis Progression According to the Findings of Transient Elastometry
Description: Decrease in liver stiffness and absence of a fibrosis progression according to the findings of transient elastometry (fibroscan) at week 24 compared to baseline
Time Frame: 24 weeks
Population: mITT
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Arm A | Arm B | Arm C | Arm D
Number analyzed (Participants) | 28 | 32 | 30 | 28
kPa
  Baseline: number analyzed (Participants) | 19 | 25 | 20 | 18
  Baseline | 14.45 (6.37) | 17.18 (11.49) | 16.00 (7.37) | 16.20 (7.83)
  Change from Baseline to Week 24: number analyzed (Participants) | 19 | 23 | 20 | 14
  Change from Baseline to Week 24 | -2.85 (2.65) | -2.52 (6.21) | -3.38 (3.83) | -0.78 (3.17)

9. Secondary Outcome: Number of Participants With Improvement of Histological Findings According to the Liver Biopsy Results
Description: Change (improvement/ worsening) in fibrosis and histological activity stage according to the liver biopsy study results at week 24 compared to baseline.
  Liver fibrosis was evaluated by histological staging systems with stage 0 corresponding to absence of fibrosis and with the highest score (the last stage in all systems) corresponding to cirrhosis.
  Improvement is defined as a decrease of at least 1 point in histological staging systems; worsening is defined as an increase of at least 1 point.
  Data should be interpreted with caution due to low number of paired biopsies available.
Time Frame: 24 weeks
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm D
Number analyzed (Participants) | 7 | 5 | 7 | 4
Participants
  Ishak fibrosis score: Improvement | 1 | 1 | 3 | 1
  Ishak fibrosis score: No change | 3 | 1 | 2 | 1
  Ishak fibrosis score: Worsening | 3 | 3 | 2 | 2
  Knodell fibrosis score: Improvement | 1 | 1 | 3 | 2
  Knodell fibrosis score: No change | 2 | 2 | 2 | 0
  Knodell fibrosis score: Worsening | 4 | 2 | 2 | 2
  Metavir fibrosis stage: Improvement | 2 | 1 | 3 | 1
  Metavir fibrosis stage: No change | 1 | 2 | 4 | 2
  Metavir fibrosis stage: Worsening | 4 | 2 | 0 | 1
  Metavir activity grade: Improvement | 2 | 2 | 3 | 3
  Metavir activity grade: No change | 4 | 1 | 3 | 0
  Metavir activity grade: Worsening | 1 | 2 | 1 | 1
  Histological activity index: Improvement | 4 | 2 | 3 | 3
  Histological activity index: No change | 0 | 1 | 1 | 0
  Histological activity index: Worsening | 3 | 2 | 3 | 1

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | Arm A | Arm B | Arm C | Arm D
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/32 | 0/30 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 3/32 | 2/30 | 1/28
Other Adverse Events (participants affected / at risk) | 18/28 | 19/32 | 21/30 | 13/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=28) | Arm B (N=32) | Arm C (N=30) | Arm D (N=28)
ALT increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=28) | Arm B (N=32) | Arm C (N=30) | Arm D (N=28)
Total bile acids increased (Investigations) | 8 (12) | 12 (20) | 15 (24) | 6 (8)
ALT increased (Investigations) | 4 (4) | 5 (9) | 9 (12) | 4 (10)
AST increased (Investigations) | 3 (3) | 7 (10) | 8 (12) | 3 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 5 (10) | 2 (5) | 3 (4)
Fatigue (General disorders) | 1 (1) | 2 (2) | 5 (6) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (4) | 3 (11) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 4 (8) | 0 (0) | 3 (4)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2) | 3 (4) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 2 (2) | 3 (3) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 4 (4) | 2 (4) | 0 (0) | 1 (1)
GGT increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Lymphopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 1 (2) | 2 (6) | 0 (0)
Amylase increased (Investigations) | 1 (1) | 1 (1) | 2 (4) | 0 (0)
Haemoglobin decreased (Investigations) | 2 (3) | 0 (0) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
INR increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Reticulocyte count decreased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Bilirubin conjugated increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ECG abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
APTT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (4) | 1 (1) | 0 (0)
Lymphocytosis (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Eosiniphilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Monocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Monocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 2 (2) | 1 (1) | 2 (3) | 0 (0)
Influenza like illness (General disorders) | 2 (4) | 1 (1) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 2 (2) | 0 (0) | 1 (2) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection sire paraesthesia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral dysaesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 2 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infected bite (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Perfume sensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Leukocyturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal variceal ligation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Menstrual disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: Protocol_v.7.0_28.09.2017_Russia + SAP + ICF (2017-09-28): https://cdn.clinicaltrials.gov/large-docs/21/NCT03546621/Prot_SAP_ICF_000.pdf
  • Study Protocol: Protocol_v.3.0_25.12.2107_Germany (2017-12-25): https://cdn.clinicaltrials.gov/large-docs/21/NCT03546621/Prot_001.pdf